CLINICAL TRIAL: NCT06367647
Title: Investigation of the Detection Rate of Pathogenic Viruses in the Feces of Individuals With Non-gastrointestinal Infections
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Yan He, Professor, Zhujiang Hospital
Other Study IDs: zhujiangjy-20240229
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Virus Infections
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- apparently healthy individuals
- parenteral virus infected patients

SUMMARY:
This project is a cross-sectional study. Investigators plan to search and collect 1600 publicly published fecal metagenomic and metatranscriptome data through the Pubmed database, by summarizing and analyzing them to construct an enterovirus database. 200 apparently healthy individuals are planned to be enrolled. At the time of enrollment, fecal specimens of participants will be collected, and their demographic characteristics, disease and medication history, gastrointestinal status, dietary habits, lifestyle habits, and mental health information will be recorded. Another 200 specimens will be collected from patients with parenteral virus infection. The demographic characteristics and pathogen test results of the parenteral virus infected patients will be reviewed and recorded. By virus metagenomic sequencing on fecal specimens, investigators will identify which viruses can be detected in the intestinal tract of apparently healthy people, and to explore whether parenteral infection viruses can be detected in feces.

ELIGIBILITY:
Inclusion Criteria:

1. age ranged from 18 to 75 years;
2. no obvious symptoms and signs of the disease;
3. not taking a drug for a long time;
4. good psychological condition ;
5. no unhealthy lifestyle;
6. willing to participate in the study, sign the informed consent, fill out the questionnaire and provide fecal samples.

Exclusion Criteria:

1. pregnant and lactating women;
2. suffering from certain diseases, such as cardiovascular disease, digestive system disease and nervous system disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparent healthy people are those who do not have clinically obvious symptoms and signs, but may have underlying health problems or premorbid conditions.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-04 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
virus infection checklist | 2024.3-2025.12
  Viral infections in the respiratory system, digestive system, urinary system, cardiovascular system, etc.

SECONDARY OUTCOMES:
general information of apparently healthy individuals by questionnaire | 2024.3-2025.12
  The general information of participants will be collected through questionnaire, which includes demographic characteristics, disease and medical history, gastrointestinal status, dietary habits, and lifestyle habits.
Self-Rating Anxiety Scale SAS | 2024.3-2025.12
  Apparently healthy individuals will fill out this scale. The total score of the scale is 25-100. The cut-off value of SAS standard score is 50 points, with 50-59 points indicating mild anxiety, 60-69 points indicating moderate anxiety, and 69 points or above indicating severe anxiety.
Self-rating depression scale SDS | 2024.3-2025.12
  Apparently healthy individuals will fill out this scale. The total score of the scale is 25-100, with 53 points indicating normal, 53-62 points indicating mild depression, 63-72 points indicating moderate depression, and above 72 points indicating severe depression.
Pittsburgh sleep quality index PSQI | 2024.3-2025.12
  Apparently healthy individuals will fill out this scale. The total score of the scale is 0-21 points and can be divided into three levels. PSQI score ≤ 4 indicates good sleep quality, PSQI score ≤ 7 indicates average sleep quality, and PSQI score ≥ 8 indicates poor sleep quality (sleep disorders). Higher PSQI total scores indicate poorer sleep quality.
demographic characteristics case information of parenteral virus infected patients | 2024.3-2025.12
  Investigators will retrospectively collect demographic characteristics and pathogen detection results of participants through case information.

CONTACTS AND LOCATIONS:
Overall Officials: Yan He, Doctor, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang hospital of southern medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No